CLINICAL TRIAL: NCT03195712
Title: Metabolically Healthy Obesity: Correlations Between BMI and Metabolic Syndrome Biomarkers in Class II and III Obesity
Brief Title: Metabolically Healthy Obesity: Correlations Between BMI and Metabolic Syndrome Biomarkers
Status: Completed | Type: Observational
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 12-048x
Record Dates: First submitted 2017-06-09; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Obesity
Keywords: BMI; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Class II and III Obesity: Patients enrolled in an outpatient weight loss program from 2010-2016.

SUMMARY:
The study team's research fills the gap in the obesity literature where BMI with a cut point of 35 is frequently used to show the association between BMI and metabolic syndrome biomarkers. The study team was unable to locate any papers that showed the association between metabolic syndrome biomarkers and BMI from 35 to 69.9, and especially graphically as this clinical team has presented.

DETAILED DESCRIPTION:
A positive association between BMI and metabolic health risk is often presented graphically as a J-shaped curve with BMI on the x-axis and the biomarker of interest on the y-axis. However, BMI is frequently presented in the literature with a cut point of 35 on the x-axis, leading to the assumption that the steep association continues beyond a BMI of 35. This presentation does not capture the metabolically healthy individual with obesity.

In the population of men and women with class II and II obesity who the clinical team studied, it was examined that the association between BMI as a continuous variable from 35 to 69.9 and metabolic syndrome biomarkers (total-, low density, and high density cholesterol, triglycerides, systolic and diastolic blood pressure, fasting blood glucose, and glycosylated hemoglobin), the study team found no evidence for a positive correlation between BMI and TC, LDL-C, TG, and FBG. And while the study team did find positive and significant correlations between BMI and HDL-C, SBP, DBP, and HgbA1C, the effect sizes were small and arguably clinically insignificant.

The study team's research fills the gap in the obesity literature where BMI with a cut point of 35 is frequently used to show the association between BMI and metabolic syndrome biomarkers. The clinical team was unable to locate any papers that showed the association between metabolic syndrome biomarkers and BMI from 35 to 69.9, and especially graphically as this clinical team has presented.

ELIGIBILITY:
Inclusion Criteria:

* BMI in the range of 35 - 69.9
* Men and Women over age 25

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: BMI 35- 69.9 Men and Women over age 25
Sampling Method: Non-Probability Sample
Enrollment: 691 (Actual)
Dates: Start 2012-09-04 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
The association between BMI from 35 - 69.9 and Total cholesterol | 7 years
  The statistical association between a range of BMIs from 35 to 69.9 kg/m2 and total cholesterol reported in mg/dl. Blood draw was performed at an independent lab as prescribed by the patients' private physician and reported to the weight loss program at Mount Sinai St. Luke's Hospital prior to the patient starting the program. To determine the association between the BMIs and total cholesterol a linear regression analysis was performed and reported graphically. The regression equation, R2, and the p-value for the regression were presented on the graph.

SECONDARY OUTCOMES:
The association between BMI from 35 - 69.9 and HDL- cholesterol | 7 years
  The statistical association between a range of BMIs from 35 to 69.9 kg/m2 and HDL-cholesterol reported in mg/dl. Blood draw was performed at an independent lab as prescribed by the patients' private physician and reported to the weight loss program at Mount Sinai St. Luke's Hospital prior to the patient starting the program. To determine the association between the BMIs and HDL-cholesterol a linear regression analysis was performed and reported graphically. The regression equation, R2, and the p-value for the regression were presented on the graph.
The association between BMI from 35 - 69.9 and LDL- cholesterol | 7 years
  The statistical association between a range of BMIs from 35 to 69.9 kg/m2 and LDL-cholesterol reported in mg/dl. Blood draw was performed at an independent lab as prescribed by the patients' private physician and reported to the weight loss program at Mount Sinai St. Luke's Hospital prior to the patient starting the program. To determine the association between the BMIs and LDL-cholesterol a linear regression analysis was performed and reported graphically. The regression equation, R2, and the p-value for the regression were presented on the graph.
The association between BMI from 35 - 69.9 and Triglycerides | 7 years
  The statistical association between a range of BMIs from 35 to 69.9 kg/m2 and triglycerides reported in mg/dl. Blood draw was performed at an independent lab as prescribed by the patients' private physician and reported to the weight loss program at Mount Sinai St. Luke's Hospital prior to the patient starting the program. To determine the association between the BMIs and triglycerides a linear regression analysis was performed and reported graphically. The regression equation, R2, and the p-value for the regression were presented on the graph.
The association between BMI from 35 - 69.9 and Systolic Blood Pressure | 7 years
  The statistical association between a range of BMIs from 35 to 69.9 kg/m2 and systolic blood pressure reported in mm/Hg. Resting blood pressure was performed by the patients' private physician at their private office and reported to the weight loss program at Mount Sinai St. Luke's Hospital prior to the patient starting the program. To determine the association between the BMIs and systolic blood pressure a linear regression analysis was performed and reported graphically. The regression equation, R2, and the p-value for the regression were presented on the graph.
The association between BMI from 35 - 69.9 and Diastolic Blood Pressure | 7 years
  The statistical association between a range of BMIs from 35 to 69.9 kg/m2 and diastolic blood pressure reported in mm/Hg. Resting blood pressure was performed by the patients' private physician at their private office and reported to the weight loss program at Mount Sinai St. Luke's Hospital prior to the patient starting the program. To determine the association between the BMIs and diastolic blood pressure a linear regression analysis was performed and reported graphically. The regression equation, R2, and the p-value for the regression were presented on the graph.
The association between BMI from 35 - 69.9 and Fasting blood glucose | 7 years
  The statistical association between a range of BMIs from 35 to 69.9 kg/m2 and fasting blood glucose reported in mg/dl. Blood draw was performed at an independent lab as prescribed by the patients' private physician and reported to the weight loss program at Mount Sinai St. Luke's Hospital prior to the patient starting the program. To determine the association between the BMIs and fasting blood glucose a linear regression analysis was performed and reported graphically. The regression equation, R2, and the p-value for the regression were presented on the graph.
The association between BMI from 35 - 69.9 and Hemoglobin A1C | 7 years
  The statistical association between a range of BMIs from 35 to 69.9 kg/m2 and hemoglobin A1C reported in percent (%). Blood draw was performed at an independent lab as prescribed by the patients' private physician and reported to the weight loss program at Mount Sinai St. Luke's Hospital prior to the patient starting the program. To determine the association between the BMIs and hemoglobin A1C a linear regression analysis was performed and reported graphically. The regression equation, R2, and the p-value for the regression were presented on the graph.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Weil, M.Ed, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai St, Luke's, New York, New York, United States